CLINICAL TRIAL: NCT06992505
Title: Assessment of Macrophage Activation syndromE in STill's Disease: Retrospective Chart Analysis of Patient hIstory, Symptom Resolution and TreAtment Characteristics in Italy (AMETISTA)
Brief Title: Assessment of Macrophage Activation syndromE in STill's Disease in Italy
Acronym: AMETISTA
Status: Completed | Type: Observational
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Other Study IDs: Sobi.EMAPALUMAB-106
Record Dates: First submitted 2025-05-09; First posted 2025-05-28 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Macrophage Activation Syndrome (MAS); Still Disease, Juvenile Onset; Still's Disease, Adult-Onset
MeSH Terms: conditions — Macrophage Activation Syndrome; Arthritis, Juvenile; Still's Disease, Adult-Onset

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assessment of macrophage activation syndrome in Still's disease:

retrospective chart analysis of patient history, symptom resolution and treatment characteristics in Italy

DETAILED DESCRIPTION:
This is an observational, retrospective cohort study on the treatment utilization and outcomes of Macrophage Activation Syndrome (MAS) refractory to glucocorticoids (GC) in patients with Still's disease. The study will be conducted entirely through medical chart abstraction; all data will be taken from the patient's medical record, with no additional assessments. The study will be conducted in Italy.

ELIGIBILITY:
Inclusion Criteria:

* Age >6 months and ≤80 years at the beginning of the index MAS episode.
* Diagnosis of Still's disease (sJIA or AOSD diagnosis).
* Diagnosis of MAS according to treating physician in the medical record.
* Patients who have received at least 3 consecutive days of GC after diagnosis of MAS and/or are judged by the Investigator to be refractory to GC due to clinical worsening of patient's condition.
* The onset of the index MAS episode occurred between 01 January 2012 and 30 September 2022.
* According to local regulations, waivers of consent will be sought for study participants from the appropriate regulatory authorities and/or the independent ethics committee (IEC)/institutional review board (IRB). o For patients not covered by waivers of consent, signed, and dated informed consent provided by the patient, or the patient's legally authorized representative(s) for patients under the legal age (with patient assent, as applicable) or who have died, should be obtained before any study-related activities are undertaken.

Exclusion Criteria:

* A diagnosis of primary HLH prior to the beginning of the index MAS episode.
* Confirmed malignancy prior to the beginning of the index MAS episode.
* Patient treated with any investigational product as a part of clinical trial during the index MAS episode.

Ages: 6 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include patients with Still's disease who were diagnosed with MAS that was refractory to GC treatment.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2025-06-06 (Actual); Primary Completion 2025-11-27 (Actual); Study Completion 2025-11-27 (Actual)

PRIMARY OUTCOMES:
Overall survival | from 2012 to 2022 (data abdstraction period)
  defined as the survival time of patients from the index date
Time to laboratory value normalization | up to 24 weeks
  defined as the time to normalization for key laboratory values
Time to MAS laboratory remission | up to 24 weeks
  defined as the time from index date to the last date of normalization of key laboratory assessments
Time to partial MAS laboratory remission | up to 24 weeks
  defined as the time from index date to the last date of normalization of at least 3 of the key laboratory assessments
Time to tapering of GCs | from index date to the last of 7 consecutive days receiving ≤1 mg/kg/day of prednisone (PDN) equivalent dose
  defined as the time from index date to the last of 7 consecutive days receiving ≤1 mg/kg/day of prednisone (PDN) equivalent dose
Number of recurrent MAS episodes | from hospital discharge or 26-weeks from the index date, whichever occurs later, until the end of study data collection]
  defined as the number of MAS episodes occurring any time after the end of the data collection period for the index MAS episode (hospital discharge or 26-weeks from the index date, whichever occurs later) until the end of study data collection
Administration of organ support care | from the index date until either the hospital discharge or 26 weeks, whichever occurs later
  defined as the proportion of patients receiving hemodialysis, assisted ventilation, cardiac support, or inotropic drugs at any time from the index date until either the hospital discharge or 26 weeks, whichever occurs later
Characteristics of MAS treatment | up to 24 weeks
  Concomitant medications
Clinical signs | at index date and 8 weeks after index date (allowed time window 6 to 12 weeks)
  Patients experiencing MAS symptoms if present (documentation in free text)

SECONDARY OUTCOMES:
Time to hospital discharge | up to 24 weeks
  defined as time from the index date to discharge from the hospital
Time to intensive care unit (ICU) discharge | up to 24 weeks
  defined as time from index date to ICU discharge
Normalization of key laboratory values | Week 8 after index date (allowed time window 6 to 12 weeks)
  Normalization of key laboratory values at Week 8 after index date (allowed time window 6 to 12 weeks)
MAS laboratory remission | at Week 8 after index date (allowed time window 6 to 12 weeks).
  Normalization of Key laboratory values at Week 8 after index date (allowed time window 6 to 12 weeks).
Partial MAS laboratory remission | at Week 8 after index date (allowed time window 6 to 12 weeks)
  Normalization of at least 3 key laboratory values at Week 8 after index date (allowed time window 6 to 12 weeks)
Duration of Clinical Response | up to 24 weeks
  defined as the time (in days) from the date of first documented MAS laboratory remission until the date of first documented occurrence of a new MAS episode as per Investigator's assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Study Physician, Study Director — Swedish Orphan Biovitrum
Locations (2):
- Italy (2):
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale Pediatrico Bambin Gesù, Rome